CLINICAL TRIAL: NCT01531023
Title: What is the Outcome of Treatment of Urinary Tract Infections Caused by Bacteria Producing Extended Spectrum Betalactamase in a Primary Care Setting?
Brief Title: Treatment of Extended Spectrum Betalactamase Producing Bacteria Causing Urinary Tract Infections in General Practice
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: University Hospital of North Norway (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); The Hospital of Vestfold (Other); Vestre Viken Hospital Trust (Other); University Hospital, Akershus (Other); Unilabs (Unknown)
Responsible Party: Principal Investigator, Marianne Bollestad, MD, University of Oslo
Other Study IDs: 2011/2214-3
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Tract Infections
Keywords: Extended-Spectrum Beta-lactamase Producing Bacteria
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urinesamples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ESBL producing E. coli bacteria: Group of patients with identified ESBL producing E.coli in a urine sample taken in a primary care setting.
- Non-ESBL E.coli urinary tract infection: E.coli bacteria found in the setting of a urinary tract infection in a primary care setting where ESBL producing bacteria are not found.

SUMMARY:
The prevalence of extended spectrum beta-lactamase (ESBL) producing bacteria found in urine sample cultures has been increasing over the past decades.

The study hypothesis is to assess the clinical and microbiological outcome of pivmecillinam treatment of ESBL producing E. coli and K. Pneumoni, as well as to observe the clinical and microbiological outcome of the same group of bacteria treated with other antiinfectious agents.

Samples are gathered in primary care setting.

ELIGIBILITY:
Inclusion Criteria:

- All patients were urinary sample taken in a primary care setting shows significant growth of ESBL producing E. coli.

Above age 16.

Exclusion Criteria:

- Sample from patients in hospital care or living in nursing home facilities. Inability to understand and sign information leaflet.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from all patients ages 16 and over who are diagnosed with an urinary tract infection where an ESBL producing bacteria (E. coli) is found. The urinary tract infection must be diagnosed and treated in a primary care setting.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of days until symptomatic resolution | Two weeks after finishing the primary antibiotic treatment
  Number of days from the start of treatment that the patient feels completely free of urinary tract symptoms Number of days after start of antibiotic treatment with mecillinam when the patient feels free of symptoms from the urinary tract

SECONDARY OUTCOMES:
Number of patients with ESBL producing bacteria detected in a urine sample taken two weeks after finishing initial treatment | Two weeks after end of initial treatment
Number of patients who received a second treatment regime in the follow-up period | 2 weeks after end of initial treatment
  Number of patients who received a secondary antibiotic treatment to obtain clinical cure.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindbaek, Md PhD, Study Director — University of Oslo
Locations (7):
- Norway (7):
  - Vestre Viken Hospital Trust, Bærum
  - University Hospital Akershus, Lørenskog
  - Unilabs, Skien
  - Helse Stavanger HF, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim
  - Vestfold Hospital Trust, Tønsberg

REFERENCES:
- [Derived] Bollestad M, Grude N, Solhaug S, Raffelsberger N, Handal N, Nilsen HS, Romstad MR, Emmert A, Tveten Y, Soraas A, Jenum PA, Jenum S, Moller-Stray J, Weme ET, Lindbaek M, Simonsen GS; (the Norwegian ESBL UTI study group). Clinical and bacteriological efficacy of pivmecillinam treatment for uncomplicated urinary tract infections caused by ESBL-producing Escherichia coli: a prospective, multicentre, observational cohort study. J Antimicrob Chemother. 2018 Sep 1;73(9):2503-2509. doi: 10.1093/jac/dky230. PMID 29982514